CLINICAL TRIAL: NCT07247630
Title: Comparison of Permethrin-Based Treatment Strategies Against Scabies in Infants and Young Children
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Shanza zafar, Doctor, Pak Emirates Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A/28/ERC.63.25
Record Dates: First submitted 2025-10-01; First posted 2025-11-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Scabies
Keywords: Permethrin based treatment strategies
MeSH Terms: conditions — Scabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard permethrin treatment (Active Comparator): Standard permethrin treatment
  Interventions: Drug: Permethrin 5%
- Intensified permethrin treatment (Active Comparator): Intensified permethrin treatment
  Interventions: Drug: Permethrin 5%

INTERVENTIONS:
Drug: Permethrin 5% — permethrin application

SUMMARY:
To compare the efficacy of different permethrin-based therapies for scabies infestations in infants and young children.

DETAILED DESCRIPTION:
Globally, Scabies infects 300 million people each year and among children of developing countries, its prevalence is estimated to be about 5-10%.In Pakistan, Scabies accounts for 38% of dermatological diseases. Males are more prone to infestation than females, and early school- aged children are the most vulnerable as it is usually transmitted by prolonged skin-skin contact.

It was more widespread in urban than in rural areas with a distinct seasonal pattern, with the biggest infestation occurring in the winter and the lowest in the summer with all risk factors accounting for 89% of the variation in its prevalence.The classic scabies symptoms include an erythematous papular eruption, burrows, and intense itching with a predilection for fingers, axilla, elbows, waist, belly, groin, genital area, etc. Several antiscabietic treatment options exist, including topically applied permethrin, benzyl benzoate (BB) and crotamiton, and oral ivermectin.5 Repeated administration of topical permethrin 5%, topical BB 10-25% or systemic ivermectin dosed at 200 μg/kg body weight is currently recommended as first-line treatment by the 2017 European guidelines for the management of scabies.Permethrin, a synthetic pyrethroid with scabicidal and ovicidal activity, disrupts the function of the voltage-gated sodium channels in the neuronal membrane of the mites, resulting in paralysis and death. Permethrin is highly effective against scabies and well- tolerated without major side-effects, as it is minimally absorbed through the skin and rapidly eliminated, thus exerting minimal systemic presence in humans.Hence, it is recommended as a first-line therapy for adults and children in many countries

ELIGIBILITY:
Inclusion Criteria:

* 1 month to 4 years age.
* Both gender
* Scabies as defined in operational definition

Exclusion Criteria:

* • Drug sensitivity test results for hypersensitivity to permethrin

  * Having renal or hepatic impairment.
  * Individuals with additional long-term skin and systemic disorders (such as diabetes, hypertension, asthma, epilepsy, acne, psoriasis)

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Treatment of scabies | 15 days
  For efficacy, we will see microscopy (presence of any one by examine skin scraping under a microscope for mites(eyeless and spherical in shape with eight legs parasite)/eggs (oval shape).The absence of these will be considered significant.

SECONDARY OUTCOMES:
Scabies | 15 days
  Absence of burrows on skin
Scabies | 15 days
  Absence of pruritus

CONTACTS AND LOCATIONS:
Locations (1):
- Pak emirates military hospital,Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No